CLINICAL TRIAL: NCT03382392
Title: Increased Resting Energy Expenditure Compared to Six Predictive Theoretical Equations in Amyotrophic Lateral Sclerosis: a Study Versus Controls
Brief Title: Hypermetabolism in ALS Using Six REE Formulas
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: mREE
Record Dates: First submitted 2017-12-13; First posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis,; Resting energy expenditure; Predictive equation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ALS
  Interventions: Other: Assesment of REE in ALS patients compared to control populations and to compare six formulas commonly used to predict REE.
- control 1
- control 2

INTERVENTIONS:
Other: Assesment of REE in ALS patients compared to control populations and to compare six formulas commonly used to predict REE.
  Groups: ALS

SUMMARY:
Introduction: About 50-60% of Amyotrophic Lateral Sclerosis (ALS) is characterized by hypermetabolism, defined as 10% or more excess resting energy expenditure (REE) compared to theoretical values. Harris and Benedict's (HB) formula is the equation mainly used to predict REE, but others are also applied in current practice. The present study aimed to assess REE in ALS patients compared to control populations and to compare six formulas commonly used to predict REE.

Nutritional assessments were performed in ALS patients and in two control populations without hypermetabolism: healthy elderly people (control 1) and patients with non-restrictive-eating disorders (control 2). Weight, height and body composition (by bioimpedance analysis) were assessed.

EE was measured (mREE) by indirect calorimetry and calculated (cREE) using HB 1919 and 1984, World Schofield, De Lorenzo, Johnstone and Mifflin formulas. Mann-Whitney and Chi2 tests were used to compare the equations.

ELIGIBILITY:
Inclusion Criteria:

* ALS patients
* 18 years old or more
* IC and nutritional assessment within 1.5 months
* delay between diagnosis and IC < 12 months

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ALS patients
Sampling Method: Non-Probability Sample
Enrollment: 449 (Actual)
Dates: Start 1996-11 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Measure of REE | indirect calorimetry (IC) and nutritional assessment within 1.5 months, and diagnosis and IC within 12 months
  EE was measured (mREE) by indirect calorimetry and calculated (cREE) using Harris and Benedict's (HB) formula

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges, France

IPD SHARING:
Plan to Share IPD: No